CLINICAL TRIAL: NCT04598191
Title: Effect of Intraoperative Iloprost Inhalant on Hemodynamic Stability in Patients Undergoing Off-pump Coronary Artery Bypass Graft Surgery: a Randomized, Blinded Clinical Trial
Brief Title: Effect of Intraoperative Iloprost Inhalant on Hemodynamic Stability in Patients Undergoing Off-pump Coronary Artery Bypass Graft Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2020-0907
Record Dates: First submitted 2020-10-12; First posted 2020-10-22 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Coronary Artery Occlusive Disease
MeSH Terms: interventions — Iloprost; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients are divided into 2 groups, who are administered aerosolized iloprost through a nebulizer connected to the inspiratory limb of the respiratory system, or who are administered same volume of normal saline at the same time and in the same manner.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants, all care providers, investigators nor outcomes assessors know the treatment allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Participants in this group are administered inhaled normal saline.
  Interventions: Drug: Control (Normal saline)
- iloprost group (Experimental): Participants in this group are administered inhaled iloprost.
  Interventions: Drug: Iloprost

INTERVENTIONS:
Drug: Iloprost — Participants in "Iloprost group" will be administered aerosolized 20 μg iloprost in 15 min through a nebulizer connected to the inspiratory limb of the respiratory system when the internal mammary artery harvesting is done.
  Arms: iloprost group
Drug: Control (Normal saline) — Participants in "Control group" will be administered aerosolized 5 ml of normal saline in 15 min through a nebulizer connected to the inspiratory limb of the respiratory system when the internal mammary artery harvesting is done.
  Arms: Control group

SUMMARY:
Considering that the cause of hemodynamic instability during OPCAB is closely related to right ventricular dysfunction with pulmonary artery hypertension, the use of inhaled iloprost (a selective pulmonary vasodilator) in patients undergoing OPCAB maybe beneficial for hemodynamic management. Previous research has showed that inhaled iloprost reduce pulmonary arterial pressure and pulmonary vascular resistance. Therefore, by administering inhaled iloprost before the graft anastomosis might improve cardiac output, mixed venous blood oxygen saturation, and pulmonary oxygenation during the surgery especially during the graft anastomosis.

The objective of our study is to evaluate the effect of inhaled Iloprost on hemodynamic stability in patients undergoing off-pump coronary artery bypass graft surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years and undergoing off-pump coronary artery bypass graft surgery with any of the following condition:
* High risk of hemodynamically unstable (patient in NYHA functional class III-IV, or mean pulmonary-artery pressure ≥ 25 mm Hg or right ventricular systolic pressure ≥ 50mmHg in preoperative echo findings, preoperative left ventricular ejection fraction < 50%, acute myocardial infarction within 1 month of surgery, ventricular fibrillation)
* History of previous cardiac operation (redo)
* Left main coronary artery disease
* Lesion at all three major coronary arteries

Exclusion Criteria:

* Emergency operation
* Patients undergoing minimally Invasive Direct Coronary Artery Bypass
* Patients with cardiogenic shock or ventricular-assist device (eg. ECMO, IABP)
* Patients with pre-existing infections prior to surgery (eg. sepsis)
* Patients with liver cirrhosis
* Patients with hemorrhagic disease / bleeding risk (history of active peptic ulcer, intracranial hemorrhage, congenital hemorrhagic disease etc.)
* Patients with cerebrovascular event (TIA, stroke) within 3 months
* Patients with symptomatic asthma/chronic obstructive pulmonary disease who are receiving treatment such as inhaler or steroid
* Patient with severe chronic kidney disease (GFR(CKD-EPI) <30ml/min/1.73m2)
* Patient with acute kidney injury
* Patients who have participated in other clinical studies that may affect prognosis
* Patients who cannot understand the informed consent (eg. Foreigner)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative cardiac index | 5 minutes before iloprost administration
  Compare the lowest intraoperative cardiac index between the Iloprost group and the control group during surgery, especially during the graft anastomosis.
Intraoperative cardiac index | 30 minutes after Iloprost administration
  Compare the lowest intraoperative cardiac index between the Iloprost group and the control group during surgery, especially during the graft anastomosis.
Intraoperative cardiac index | 5 minutes after the start of graft anastomosis
  Compare the lowest intraoperative cardiac index between the Iloprost group and the control group during surgery, especially during the graft anastomosis.
Intraoperative cardiac index | 5 minutes after pericardial closure
  Compare the lowest intraoperative cardiac index between the Iloprost group and the control group during surgery, especially during the graft anastomosis.

SECONDARY OUTCOMES:
systemic arterial blood pressure for the intraoperative hemodynamic parameters | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure
central venous pressure(CVP in mmhg) for the intraoperative hemodynamic parameters | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure
pulmonary artery pressure for the intraoperative hemodynamic parameters | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure
heart rate for the intraoperative hemodynamic parameters | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure
EKG rhythm for the intraoperative hemodynamic parameters | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure
mixed venous oxygen saturation for the intraoperative hemodynamic parameters | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure
PaO2/FiO2 ratio for the ventilation and oxygenation parameter | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure
oxygen saturation in arterial blood for the ventilation and oxygenation parameter | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure
arterial blood gas (ABG) test for oxygenation parameter | 15 minutes after induction of anesthesia (baseline), 30 minutes after Iloprost administration, 5 minutes after pericardial closure
airway pressure (peak, plateau, PEEP) for the lung mechanics | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure
dynamic compliance for the lung mechanics | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure
driving pressure for the lung mechanics | 15 minutes after induction of anesthesia (baseline), 5 minutes before iloprost administration, 30 minutes after Iloprost administration, 5 minutes after the start of graft anastomosis, 5 minutes after pericardial closure

CONTACTS AND LOCATIONS:
Overall Officials: Jae Kwang Shim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko SH, Shim JK, Song JW, Soh S, Kwak YL. Inhaled iloprost in off-pump coronary artery bypass surgery: a randomized controlled trial. Can J Anaesth. 2024 Apr;71(4):479-489. doi: 10.1007/s12630-023-02672-3. Epub 2023 Dec 26. PMID 38148468